CLINICAL TRIAL: NCT01794455
Title: Effects of Cerebral Hypoperfusion and Its Reversal on Late-Life Depression
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment difficulties
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Warren Taylor, Associate Professor of Psychiatry, Vanderbilt University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VR5642
Record Dates: First submitted 2013-02-12; First posted 2013-02-18 (Estimated); Results first posted 2016-10-20 (Estimated); Last update posted 2016-10-20 (Estimated); Status verified 2016-08

CONDITIONS: Depression; Hypertension
Keywords: Depression; Depressive Disorder; Geriatrics; Hypertension
MeSH Terms: conditions — Depression; Hypertension; Depressive Disorder | interventions — Sertraline; candesartan; candesartan cilexetil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Phase 1: Sertraline (Experimental): Eight-week trial of sertraline mono therapy, dosing ranging from 50mg- 200mg daily.
  Interventions: Drug: Sertraline
- Phase 2: Candesartan (Experimental): For subjects who do not remit to sertraline, they will receive candesartan for 12 weeks, with doses ranging from 4mg - 32mg daily.
  Interventions: Drug: Candesartan

INTERVENTIONS:
Drug: Sertraline — 50mg - 200mg daily
  Other Names: Zoloft
  Arms: Phase 1: Sertraline
Drug: Candesartan — 4mg - 32mg daily
  Other Names: Atacand
  Arms: Phase 2: Candesartan

SUMMARY:
This pilot proposal will test the hypothesis that altered cerebral vessel reactivity and cerebral hypoperfusion (decreased blood flow to the brain) is a core mechanism underlying the relationship between vascular disease and depression in older adults. The long-term objective of this line of research is to: A) determine the relationship between vascular reactivity, cerebral hypoperfusion and the persistence of late-life depression and B) determine if improving cerebral perfusion with angiotensin receptor blockers (ARBs) improves depression outcomes.

DETAILED DESCRIPTION:
This study will examine how magnetic resonance imaging (MRI) measures of cerebral perfusion relate to antidepressant response. There are two phases to the study. In the first phase, we will examine how cerebral perfusion is related to response to sertraline, a commonly used antidepressant. In the second phase, we will examine individuals who do not respond to sertraline or other selective serotonin reuptake inhibitors (SSRI). We will examine if candesartan, an ARB, improves depression and if it does so by improving cerebral perfusion.

After providing informed consent, participants will undergo medical and psychiatric screening. Participants determined to be eligible at the screen will proceed to a baseline evaluation, which will include brief cognitive neuropsychological testing and MRI. Participants will then begin open-label sertraline for eight weeks (baseline to week 8). Dosing will begin at 50mg daily and, based on response and tolerability, can increase up to the FDA approved maximum dose of 200mg daily.

After the eight weeks, participants will be re-evaluated and complete another MRI. Those who respond to sertraline and experience remission of their depression will end their study participation. Those who do not experience remission will continue to the phase 2 open-label candesartan arm.

The candesartan arm will last for 12 weeks (week 8 to week 20). Dosing will begin at 4mg daily and can increase to a maximum dose of 32mg, based on tolerability and response. Participants will be monitored closely, and other antihypertensive medications adjusted to avoid low blood pressure. At the end of the 12-week trial, participants will again complete MRI and neuropsychological testing. Their study participation will then end.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 years or older
2. Diagnosis of Major Depressive Disorder, single or recurrent episode, without psychotic features by Diagnostic and Statistical Manual IV Text Revision (DSMIV-TR) criteria
3. Presence of hypertension (defined as systolic > 140 or diastolic > 90 or currently receiving antihypertensive therapy)
4. Minimum depression severity of ≥ 15 on the Montgomery-Asberg Depression Rating Scale (MADRS)
5. Cognitively intact or with mild cognitive deficits, with a minimum score ≥ 23 on the Montreal Cognitive Assessment (MoCA).

Exclusion Criteria:

1. Other psychiatric Axis I disorders
2. Acute suicidality
3. Electroconvulsive therapy in the last 6 months
4. Primary neurological disorder, including dementia and stroke
5. Significant cardiovascular disease, specifically diagnosis of congestive heart failure, known bilateral renal artery stenosis, symptomatic hypotension, or critical aortic or mitral stenosis
6. Myocardial infarction or open-heart surgery in last 6 weeks
7. Serum creatinine ≥ 265 micromol /L
8. Serum potassium ≥ 5.5 mmol/L
9. MRI contraindications
10. Known allergy to sertraline or candesartan specifically or known allergy to other SSRIs or ARBs.
11. History of prolonged (> 3 weeks) or self-described severe discontinuation syndrome in the past after stopping an antidepressant.
12. Current use of an angiotensin receptor blocker
13. Current or planned psychotherapy
14. Need for continuous oxygen use or any medical disorder where the hypercapnia challenge would be contraindicated or put the subject at increased risk. This would include acute respiratory disease, chronic angina, or other unstable cardiac conditions.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren D Taylor, MD, MHSc, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Psychiatric Hospital, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Phase 1: Sertraline | Phase 2: Candesartan
Started | 0 | 1
Completed | 0 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Sertraline | Phase 2: Candesartan | Total
Number analyzed (Participants) | 0 | 1 | 1
Age, Categorical [Number; unit: participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 0 | 0
  >=65 years |  | 1 | 1
Age, Continuous [Mean (Full Range); unit: years] |  | 67 [67 to 67] | 67 [67 to 67]
Gender [Number; unit: participants]
  Female |  | 0 | 0
  Male |  | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States |  | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: MRI Arterial Spin Labeling
Description: MRI arterial spin labeling is a noninvasive approach to measuring cerebral blood flow. This relates to the Phase 1 sertraline arm.
Time Frame: Change in perfusion from baseline to week 8
Population: Could not complete MRI.
Arm/Group | Phase 1: Sertraline | Phase 2: Candesartan
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Montgomery Asberg Depression Rating Scale (MADRS)
Description: MADRS is a measure of depression severity. This outcome applies to the sertraline Phase 1 arm.
Time Frame: Week 8
Arm/Group | Phase 1: Sertraline | Phase 2: Candesartan
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quick Inventory of Depressive Symptoms, Self-Rated (QIDS-SR16)
Description: Self-report measure of depression severity. This applies to the sertraline Phase 1 arm.
Time Frame: Week 8
Arm/Group | Phase 1: Sertraline | Phase 2: Candesartan
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Quick Inventory of Depressive Symptoms, Self-Rated (QIDS-SR16)
Description: Self-report measure of depression severity (range 0 - 27, higher scores indicate more severe depressive symptoms). This applies to the candesartan Phase 2 arm.
Time Frame: Week 20
Measure: Number; unit: units on a scale
Arm/Group | Phase 1: Sertraline | Phase 2: Candesartan
Number analyzed (Participants) | 0 | 1
units on a scale |  | 11

5. Secondary Outcome: Montgomery-Asberg Depression Rating Scale
Description: MADRS is a measure of depression severity (range 0 - 60, higher scores indicate more severe depressive symptoms). This outcome applies to the candesartan Phase 2 arm.
Time Frame: Week 20
Measure: Number; unit: units on a scale
Arm/Group | Phase 1: Sertraline | Phase 2: Candesartan
Number analyzed (Participants) | 0 | 1
units on a scale |  | 22

6. Secondary Outcome: MRI Arterial Spin Labeling
Description: MRI arterial spin labeling is a noninvasive approach to measuring cerebral blood flow. This relates to the Phase 2 candesartan arm.
Time Frame: Change from week 8 to week 20
Population: MRI data could not be obtained on the one study participant due to MRI contraindications.
Arm/Group | Phase 1: Sertraline | Phase 2: Candesartan
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Phase 1: Sertraline | Phase 2: Candesartan
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Sertraline (N=0) | Phase 2: Candesartan (N=1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was ended early due to difficulty with subject recruitment. MRI data could not be obtained on that one individual due to MRI contraindications.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes